CLINICAL TRIAL: NCT02565290
Title: Effect of Mother's Supplementation Omega-3 in the Dynamics of Fetal Ductus Arteriosus: a Randomized Clinical Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple
Other Study IDs: UP4989/2014
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Pregnancy
Keywords: polyunsaturated fatty acid; fetal ductus arteriosus; inflammation
MeSH Terms: conditions — Inflammation | interventions — Docosahexaenoic Acids; Soybean Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 (Active Comparator): 2 capsules of omega 3 - 2 times a day
  Interventions: Dietary Supplement: Omega 3
- Soy oil (Placebo Comparator): 2 capsules of soy oil - 2 times a day
  Interventions: Dietary Supplement: Soy Oil

INTERVENTIONS:
Dietary Supplement: Omega 3 — Pregnant women should take 2 capsules of omega 3 (1g), 2 times a day, for 21 days.
  Arms: Omega-3
Dietary Supplement: Soy Oil — Pregnant women should take 2 capsules of placebo 3 - soy oil oil (1g), 2 times a day, for 21 days.
  Arms: Soy oil

SUMMARY:
The effect of anti-inflammatory substances on the dynamics of the fetal ductus arteriosus is well documented, but the anti-inflammatory property of polyunsaturated fatty acid omega-3 about changing this dynamic is not established. This study evaluate the relationship between supplementation of omega-3 in the dynamics of the fetal ductus arteriosus in the third trimester. Women with gestational between 28 to 32 weeks will receive capsules of omega-3 or placebo, to be consumed daily for 3 weeks.

DETAILED DESCRIPTION:
The omega-3 features similar the statins to be antioxidants and anti-inflammatory drugs and their derivatives have the function of slowing the neuro-inflammation, oxidative stress and apoptotic cell death anti-inflammatory properties. Also, they have antithrombotic effects, being related to prevent disease. Studies show that supplementation with omega-3 has a positive impact on several outcomes like cardiovascular disease, asthma, rheumatoid arthritis and Alzehimer. Objective: Evaluate the relationship between supplementation of omega-3 in the dynamics of the fetal ductus arteriosus in the third trimester. Methodology: randomized double blind clinical trial. Women with gestational age between 28 to 32 weeks, literate, over 18 years will be invited. Pregnant women with anti-inflammatory drugs, they have a higher intake of dietary polyphenols to 127mg / day or using drugs that may interfere with the absorption of omega-3 are excluded. The selected women will be randomized to receive capsules of omega-3 or placebo, to be consumed daily for 3 weeks. In the first interview, and after 3 weeks, they will respond the Questionnaire Food Frequency (QFF) to quantify polyphenols and omega 3 in their diet, weight and height will be measured and the examination of fetal echocardiography is performed.

ELIGIBILITY:
Inclusion Criteria: Women between 28 - 32 weeks pregnancy who accept participate in the study.

-

Exclusion Criteria: hypertensive , diabetic , who use anti-inflammatory drugs , HIV positive , do not take mate, black or green tea, had inflammation in the last 5 days, allergic to fish or soy.

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Pulsatility index of fetal ductus arteriosus | 28 to 32 weeks of pregnancy
  The measure will be collected before and after 21 days of supplementation with omega 3 capsules

SECONDARY OUTCOMES:
Systolic and diastolic velocity of fetal ductus arteriosus | 28 to 32 weeks of pregnancy
  The measure will be collected before and after 21 days of supplementation with omega 3
Inflammatory biomarkers (interleukins, prostaglandins, cyclooxygenase) | 28 to 32 weeks of pregnancy
  Will be collected blood before and after 21 days of supplementation with omega 3
Biomarkers of oxidative stress | 28 to 32 weeks of pregnancy
  Will be collected blood before and after 21 days of supplementation with omega 3

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Zielinsky, Doctor, Study Director — Instituto de Cardiologia do Rio Grande do Sul
Locations (1):
- Paulo Zielinsky, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Result] Zielinsky P, Piccoli AL Jr, Vian I, Zilio AM, Naujorks AA, Nicoloso LH, Barbisan CW, Busato S, Lopes M, Klein C. Maternal restriction of polyphenols and fetal ductal dynamics in normal pregnancy: an open clinical trial. Arq Bras Cardiol. 2013 Sep;101(3):217-25. doi: 10.5935/abc.20130166. Epub 2013 Aug 14. PMID 23949325
- [Result] Vian I, Zielinsky P, Zilio AM, Mello A, Lazzeri B, Oliveira A, Lampert KV, Piccoli A, Nicoloso LH, Bubols GB, Garcia SC. Development and validation of a food frequency questionnaire for consumption of polyphenol-rich foods in pregnant women. Matern Child Nutr. 2015 Oct;11(4):511-24. doi: 10.1111/mcn.12025. Epub 2013 Jan 15. PMID 23316751
- [Result] Zielinsky P, Manica JL, Piccoli AL Jr, Nicoloso LH, Barra M, Alievi MM, Vian I, Zilio A, Pizzato PE, Silva JS, Bender LP, Pizzato M, Menezes HS, Garcia SC. Fetal ductal constriction caused by maternal ingestion of green tea in late pregnancy: an experimental study. Prenat Diagn. 2012 Oct;32(10):921-6. doi: 10.1002/pd.3933. Epub 2012 Jul 23. PMID 22821626
- [Result] Bubols GB, Zielinsky P, Piccoli AL Jr, Nicoloso LH, Vian I, Moro AM, Charao MF, Brucker N, Bulcao RP, Nascimento SN, Baierle M, Alievi MM, Moresco RN, Markoski M, Garcia SC. Nitric oxide and reactive species are modulated in the polyphenol-induced ductus arteriosus constriction in pregnant sheep. Prenat Diagn. 2014 Dec;34(13):1268-76. doi: 10.1002/pd.4463. Epub 2014 Aug 22. PMID 25043716